CLINICAL TRIAL: NCT03435731
Title: Dual Obstructive Sleep Apnea (OSA) Therapy (MAS With PAP)
Brief Title: Dual Obstructive Sleep Apnea Therapy
Acronym: DOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of British Columbia (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Fernanda Almeida, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H18-00175; FCRC1801 (Other: Frontier Clinical Research Centre)
Record Dates: First submitted 2018-02-08; First posted 2018-02-19 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; Continous Positive Airway Pressure (CPAP); Mandibular Advancement Split (MAS); Mandibular Advancement Oral Appliance; Dual Therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): This group will undergo 1 month Dual Therapy.
  Interventions: Combination Product: Dual Therapy

INTERVENTIONS:
Combination Product: Dual Therapy — Concomitant use of Continuous Positive Airway Pressure (CPAP) and Mandibular Advancement Splint (MAS) therapeutic devices.

SUMMARY:
Continuous positive airway pressure (CPAP) is considered the gold standard therapy for obstructive sleep apnea (OSA). However, CPAP users sometimes experience pressure-related discomfort. It is thought that lower CPAP pressure may increase comfort and lead to greater treatment adherence.

Mandibular advancement splint (MAS) therapy has been shown to be the preferred OSA treatment option among patients. However, MAS therapy is only partially effective in some OSA patients, especially in severe cases.

It is thought that a combination of MAS and PAP therapy may benefit patients in which MAS alone is only partially effective. Using MAS and PAP at the same time is called "Dual Therapy". Dual Therapy may allow a lower CPAP pressure to be applied, which may increase patient comfort and therefore increase treatment adherence and overall effectiveness.

This study will evaluate the effectiveness of 1 month of Dual Therapy in 30 OSA patients.

DETAILED DESCRIPTION:
This is a prospective clinical trial assessing the effect of 1-month of dual therapy on patients with varying baseline OSA severity (mild to severe) who have been previously fully titrated to both PAP and MAS.

This study will be conducted at 2 research centers; the Faculty of Dentistry, University of British Columbia (UBC), Vancouver and at the Faculty of Dentistry, Université de Montréal (UdM), Montréal.

The research team will access participants' records to confirm eligibility for dual therapy. The clinical research coordinator will contact eligible patients via phone to ask if they are interested in taking part in the study. Eligible patients will also be asked if they are interested in taking part in the study during routine clinic visits. Where possible, patients will not be approached by their primary caregiver regarding participation in this study, to ensure patients do not feel pressurized into participating. Choosing not to take part in the study will not affect the participants' quality of care. If a patient is interested in taking part in the study they will be invited to review and sign the informed consent form.

Consenting participants will be asked to use both MAS and PAP (dual therapy) together for a period of 1 month. During the first week of the dual therapy, PAP pressure will be adjusted automatically for a 1-week period, after which the pressure will be set remotely by the Respiratory Therapist at the 90th percentile.

With permission, the research team will access the Sleep Apnea Dental Clinic records to collect data relating to previous treatment with MAS and PAP monotherapies. Data collected includes: PAP pressure, treatment adherence, subjective treatment assessment, Epworth Sleepiness Scale (ESS) and Functional Outcomes of Sleep Questionnaires (FOSQ), weight, blood pressure and oximetry data.

At the end of the 1-month, a subjective and objective assessment will be conducted. Subjective data will be collected using a short questionnaire that will be completed by the participants pertaining to their experience with the dual therapy in addition to completing a short term medical/treatment update form. Participants' weight and blood pressure will also be reassessed. Objective adherence will be analyzed via data obtained from the PAP modem and from DentiTrac® smart chips embedded in the MAS. OSA-related quality of life will be reassessed using ESS and FOSQ questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-80 years old who are able to freely provide informed consent;
* Prior participation in the CHOICE study;
* Have been optimally titrated to PAP and MAS therapy;
* Have both PAP and MAS appliances at home and ready for use;
* Body mass index (BMI) of 35 or less;
* ≥ 8 teeth per arch to support treatment with MAS;
* Have an objective of diagnosis of OSA based on the following criteria:
* - an Apnea-Hypopnea Index (AHI) within the range 10 ≤ AHI ≤ 70 documented with polysomnography in the last 2 years; ***OR***
* - a Respiratory Disturbance Index (RDI) within the range 20 ≤ RDI ≤ 70 documented with level III portable sleep test; ***OR***
* - an Oxygen Desaturation Index (ODI) ≥ 10;
* Sleep investigations confirming the object diagnosis of OSA have been performed within the past 4 years

Exclusion Criteria:

* Use of a full face mask as the PAP interface;
* Extensive periodontal disease with significant tooth mobility;
* Inability to protrude jaw;
* Insufficient vertical opening to accommodate treatment with MAS;
* Uncontrolled congestive heart failure (defined as a prior clinical diagnosis, an ejection cut-off of 40% or clinical sign in the opinion of a primary care physician or cardiologist) that makes it unsafe in the opinion of the investigators for the subject to participate in the trial;
* Coronary artery disease unless stable for at least 6 months and considered by the investigators to have a stable disease;
* Any history of angina, myocardial infarction or stroke;
* Any history of major depressive disorder along with current moderate-severe disease;
* Active cancer management (unless in remission for more than 1 year);
* Known renal failure (with need for dialysis);
* History of a near miss or prior automobile accident due to sleepiness within the past 12 months;
* At nighttime, 30% of the night is at ≤ 90% oxygen saturation levels.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-08 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in CPAP Pressure | Baseline (from previous treatment with CPAP) and 1 month after commencing Dual Therapy treatment.
  Optimal CPAP Pressure determined by the Respiratory Therapist (cmH2O)
Comfort | Baseline (from previous treatment) and 1 month after commencing Dual Therapy treatment.
  A subjective assessment of the Dual Therapy treatment, reported via a questionnaire.
Treatment Adherence (hrs/night) | The duration of Dual Therapy treatment (1 month).
  Adherence measured in hours per night.
Treatment Adherence (% nights) | The duration of Dual Therapy treatment (1 month).
  Adherence measured in percentage of nights of use.

SECONDARY OUTCOMES:
Daytime Sleepiness | Baseline (from previous treatment) and 1 month after commencing Dual Therapy treatment.
  Evaluation of OSA specific fatigue using Epworth Sleepiness Scale (ESS) questionnaire. ESS measures daytime sleepiness via 8 questions that ask about daytime sleepiness during common everyday conditions. The potential range of scores for any questions is from 0 to 3. Higher values represent worse outcomes. Their are no subscales for ESS. The answers to the questions are all summed up. Total score ranges between 0 and 24. A score above 10 indicates daytime sleepiness with higher scores indicating more sleepiness.
Quality of Life using Functional Outcomes of Sleep Questionnaire (FOSQ-10) | Baseline (from previous treatment) and 1 month after commencing Dual Therapy treatment.
  FOSQ-10 measures functional status and difficulty in performing everyday activities via 10 questions. The range of scores for any question is from 1 to 4. There is also a 0 score option for participants who do not engage in a particular activity for other reasons, in which case the question will be excluded. There are 5 subscales that measure: general productivity, activity level, vigilance, social outcomes, and intimacy and sexual relationships. To obtain the total score, a mean-weighted item score is computed for those subscales with more than one item. To calculate a mean-weighted item score calculate the mean of the answered items with responses > 1 for each subscale. The total score is then derived by calculating the mean of the subscale scores and multiplying that mean by five. Total score ranges between 5 and 20. Higher scores indicate better functional status.
Efficacy - Oxygen Desaturation Index | Baseline (from previous treatment) and 1 month after commencing Dual Therapy treatment.
  The number of times per hour of sleep that the blood's oxygen level drop below 97% oxygen saturation.
Efficacy - Time below 90% Saturation | Baseline (from previous treatment) and 1 month after commencing Dual Therapy treatment.
  Percentage of time during sleep that the patient's blood oxygen levels fall below 90% saturation.
Efficacy - Minimum Saturation | Baseline (from previous treatment) and 1 month after commencing Dual Therapy treatment.
  The lowest percentage saturation of the patient's blood oxygen levels during sleep.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - Université de Montréal, Montreal, Quebec